CLINICAL TRIAL: NCT01672632
Title: Fat Cell Size and Overfeeding and Etopic Study
Acronym: EAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Eric Ravussin, Principal Investigator, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PBRC 26040; 5R01DK060412 (NIH)
Record Dates: First submitted 2012-08-20; First posted 2012-08-27 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Over Eating
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Overfeeding (Experimental): We overfed 40 young, healthy adults by 40% of their baseline energy requirements for 8 weeks. The diet consisted of 41% carbohydrate, 44% fat, and 15% protein.
  Interventions: Other: Overfeeding

INTERVENTIONS:
Other: Overfeeding — We overfed 40 young, healthy adults by 40% of their baseline energy requirements for 8 weeks. The diet consisted of 41% carbohydrate, 44% fat, and 15% protein.

SUMMARY:
It has been shown that large fat cells are associated with more risks for insulin resistance and more cardiovascular risk factors such as high cholesterol or triglycerides.

DETAILED DESCRIPTION:
This study will look at fat cell size and how it affects fat deposition, insulin resistance and muscle oxidative capacity. A comparison will be made with the differences between participants with larger versus smaller fat cells in insulin resistance and blood levels of lipids. The study will also determine if characteristics of fat cells and muscle can predict the development of weight gain-induced insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Your Body Mass Index (height to weight ratio) is 22.5 to 32.5 (inclusive).
* You are 18-40 years of age.
* You are willing to enroll in an 8 week overfeeding study causing a 5-8 % weight gain.
* You are willing to eat all your meals from Pennington and only meals from Pennington for approximately 10 weeks total, even when you are full. Prior to overfeeding 2 Meals per day will be served at Pennington with lunch packed for at least 7 days. After that time participants will receive and eat all (overfeeding) meals at PBRC for 8 weeks. Post-overfeeding will consists of weight-maintenance diet for 1 week. All meals will be monitored at Pennington.
* You are willing to maintain the same level of exercise after enrollment in the study throughout the length of the study.
* You are willing to complete nutritional and activity questionnaires.

Exclusion Criteria:

* You weight > 300 lbs
* You have a history of cardiovascular disease or diabetes.
* You have a fasting blood glucose > 110 mg/dL.
* You have an average screening blood pressure > 140/90.
* You have liver disease.
* You have thyroid disease.
* Have Acid Reflux
* Had cancer in the last 5 years (Some skin cancers OK)
* Have HIV
* Have had an Eating Disorders
* You are pregnant or breastfeeding.
* You have gained or lost more than 3kg in the last 3 months
* You require chronic use of medications including diuretics, steroids and adrenergic-stimulating agents.
* You or a member of your family has a history of blood clots (deep vein thrombosis or pulmonary embolism)
* You have poor circulation, history of bypass operation in your legs, blood coagulation disorders, diagnosed peripheral arterial or vascular disease, cramping pain in your leg muscle during exercise or nerve damage to your legs
* You have varicose veins (per discretion of MD or NP)
* You have had previous GI surgery, obstructive disease of the GI tract, hyper motility disorder or a history of problems of impairment of the gag reflex.
* You have emotional problems such as clinical depression or other diagnosed psychological conditions.
* You are claustrophobic.
* You have metal objects in your body such as implanted rods or surgical clips or magnetic objects that are incompatible with the MRI/MRS.
* You smoke or use tobacco products

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Determine the effect of 8-weeks 40% high fat overfeeding in 40 healthy, young adults on adipose and skeletal muscle characteristics, ectopic fat accumulation, insulin sensitivity, and metabolic flexibility. | 10 months
  This study will investigate how fat cell size (independent of total fat mass) affects metabolic outcomes of overfeeding, including changes in fat deposition, insulin sensitivity and muscle oxidative capacity. It has been shown that large fat cells relative to fat mass are associated with higher risks for insulin resistance and type 2 diabetes.

SECONDARY OUTCOMES:
Fat Deposition | 10 Months
  Viewing of adipose tissue or body fat and skeletal muscle characteristics over a period.
Insulin Sensitivity | 10 months
  Measure and monitor the natural hormone insulin becomes less effective at lowering blood sugars. The resulting increase in blood glucose may raise levels outside the normal range and cause adverse heealth effects, depending on dietary conditions or sensitivity of cells to insulin.
Muscle Oxidative Capacity | 10 Months
  A measure of a muscle's maximal capacity to use oxygen in microliters of oxygen consumed per gram of muscle per hour.
Circadian Blood Pressure variability | 10 Months
  Blood pressure and heart rate measurement: An automatic BP monitoring device (Mortara® Ambulo 2400) for ambulatory use was attached to a BP cuff to obtain blood pressure (BP) and heart rate (HR) readings at 30-min intervals during the day (6:30 AM to 9:30 PM) and 60-min intervals at night (10 PM to 6 AM) while the participants went about their activities. Data were downloaded into the database at the end of the 7-day recording span for a chronobiological analysis. This was done at baseline, post-overfeeding and at 3 months.
Resting Endothelial function testing | 10 Months
  Endothelial function testing: Assessment of resting endothelial function was done with the participant in a fasting state, after having avoided stimulants (caffeine, tobacco, alcohol, exercise) for 12 hours, at the same fixed clock hour (range 8-10 AM), using the EndoPAT 2000 device manufactured by ITAMAR Medical®.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Ravussin, PhD, Principal Investigator — Pennington Biomedical Research Center; Alok Gupta, MD, Principal Investigator — Pennington Biomedial Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] White U, Beyl RA, Ravussin E. A higher proportion of small adipocytes is associated with increased visceral and ectopic lipid accumulation during weight gain in response to overfeeding in men. Int J Obes (Lond). 2022 Aug;46(8):1560-1563. doi: 10.1038/s41366-022-01150-y. Epub 2022 May 23. PMID 35599261
- [Derived] Hochsmann C, Fearnbach N, Dorling JL, Myers CA, Zhang D, Apolzan JW, Stewart TM, Bray GA, Ravussin E, Martin CK. Effect of 8 weeks of supervised overfeeding on eating attitudes and behaviors, eating disorder symptoms, and body image: Results from the PROOF and EAT studies. Eat Behav. 2021 Dec;43:101570. doi: 10.1016/j.eatbeh.2021.101570. Epub 2021 Oct 1. PMID 34655863
- [Derived] Johannsen DL, Marlatt KL, Conley KE, Smith SR, Ravussin E. Metabolic adaptation is not observed after 8 weeks of overfeeding but energy expenditure variability is associated with weight recovery. Am J Clin Nutr. 2019 Oct 1;110(4):805-813. doi: 10.1093/ajcn/nqz108. PMID 31204775
- [Derived] Broskey NT, Obanda DN, Burton JH, Cefalu WT, Ravussin E. Skeletal muscle ceramides and daily fat oxidation in obesity and diabetes. Metabolism. 2018 May;82:118-123. doi: 10.1016/j.metabol.2017.12.012. Epub 2018 Jan 4. PMID 29307520
- [Derived] Toledo FGS, Johannsen DL, Covington JD, Bajpeyi S, Goodpaster B, Conley KE, Ravussin E. Impact of prolonged overfeeding on skeletal muscle mitochondria in healthy individuals. Diabetologia. 2018 Feb;61(2):466-475. doi: 10.1007/s00125-017-4496-8. Epub 2017 Nov 17. PMID 29150696
- [Derived] Covington JD, Johannsen DL, Coen PM, Burk DH, Obanda DN, Ebenezer PJ, Tam CS, Goodpaster BH, Ravussin E, Bajpeyi S. Intramyocellular Lipid Droplet Size Rather Than Total Lipid Content is Related to Insulin Sensitivity After 8 Weeks of Overfeeding. Obesity (Silver Spring). 2017 Dec;25(12):2079-2087. doi: 10.1002/oby.21980. Epub 2017 Oct 25. PMID 29071793
- [Derived] Heymsfield SB, Peterson CM, Thomas DM, Hirezi M, Zhang B, Smith S, Bray G, Redman L. Establishing energy requirements for body weight maintenance: validation of an intake-balance method. BMC Res Notes. 2017 Jun 26;10(1):220. doi: 10.1186/s13104-017-2546-4. PMID 28651559
- [Derived] Peterson CM, Orooji M, Johnson DN, Naraghi-Pour M, Ravussin E. Brown adipose tissue does not seem to mediate metabolic adaptation to overfeeding in men. Obesity (Silver Spring). 2017 Mar;25(3):502-505. doi: 10.1002/oby.21721. Epub 2017 Jan 24. PMID 28117556
- [Derived] Covington JD, Noland RC, Hebert RC, Masinter BS, Smith SR, Rustan AC, Ravussin E, Bajpeyi S. Perilipin 3 Differentially Regulates Skeletal Muscle Lipid Oxidation in Active, Sedentary, and Type 2 Diabetic Males. J Clin Endocrinol Metab. 2015 Oct;100(10):3683-92. doi: 10.1210/JC.2014-4125. Epub 2015 Jul 14. PMID 26171795
- [Derived] Gilmore LA, Ravussin E, Bray GA, Han H, Redman LM. An objective estimate of energy intake during weight gain using the intake-balance method. Am J Clin Nutr. 2014 Sep;100(3):806-12. doi: 10.3945/ajcn.114.087122. Epub 2014 Jul 23. PMID 25057153
- [Derived] Johannsen DL, Tchoukalova Y, Tam CS, Covington JD, Xie W, Schwarz JM, Bajpeyi S, Ravussin E. Effect of 8 weeks of overfeeding on ectopic fat deposition and insulin sensitivity: testing the "adipose tissue expandability" hypothesis. Diabetes Care. 2014 Oct;37(10):2789-97. doi: 10.2337/dc14-0761. Epub 2014 Jul 10. PMID 25011943
- [Derived] Lam YY, Redman LM, Smith SR, Bray GA, Greenway FL, Johannsen D, Ravussin E. Determinants of sedentary 24-h energy expenditure: equations for energy prescription and adjustment in a respiratory chamber. Am J Clin Nutr. 2014 Apr;99(4):834-42. doi: 10.3945/ajcn.113.079566. Epub 2014 Feb 5. PMID 24500151